## STATISTICAL ANALYSIS PLAN

NCT Number: NCT04198363

Study Title: A Randomized Double-Blind, Phase 3 Study to Evaluate the

Efficacy and Safety of Bismuth-Containing Quadruple Therapy With Oral TAK-438 20 mg Compared to Esomeprazole 20 mg Twice Daily in Subjects With Helicobacter Pylori Infection

Study Number: Vonoprazan-3002

SAP Version and Date:

Version 3.0: 31-August-2021



#### STATISTICAL ANALYSIS PLAN

STUDY NUMBER: Vonoprazan-3002

licable Terms of Use A Randomized Double-Blind, Phase 3 Study to Evaluate the Efficacy and Safety of Bismuth-Containing Quadruple Therapy With Oral TAK-438 20 mg Compared to Esomeprazole 20 mg Twice Daily in Subjects With Helicobacter Pylori Infection

#### PHASE 3

Version: 3

Date: 24 August 2021

Prepared by:

Based on:

Biostatistics

Biostatistics Protocol Version: Amendment 03 Protocol Date: 20 October 2020

Probably of Takeda: For non-commercial use only and subject to the applicable Terms of the property of takeda: For non-commercial use only and subject to the applicable of takeda: For non-commercial use only and takeda: For non-commercial use

# 2.0 TABLE OF CONTENTS

| 1.0 TITLE PAGE | 1 |
|-----------------------------------------------------------------|-----|
| 1.1 Approval Signatures | 2 |
| 2.0 TABLE OF CONTENTS | |
| List of In-Text Tables | |
| T'A CI TE AE' | 4 |
| 3.0 LIST OF ABBREVIATIONS | 5 |
| List of in-Text Figures 3.0 LIST OF ABBREVIATIONS | 6 |
| 4.1 Primary Objective | 6 |
| 4.2 Secondary Objectives | 6 |
| 4.3 Additional Objectives | 6 |
| 4.4 Study Design | 6 |
| 5.0 ANALYSIS ENDPOINTS | 8 |
| 6.0 DETERMINATION OF SAMPLE SIZE | 9 |
| 7.0 METHODS OF ANALYSIS AND PRESENTATION | 10 |
| 7.1 General Principles | 10 |
| 7.1.1 Study Definitions | 10 |
| 7.1.2 Definition of Study Days | 11 |
| 7.1.3 Definition of Study Visit Windows | 11 |
| 7.1.4 Significance Level and Confidence Coefficient | 12 |
| 7.1.5 Conventions for Missing Adverse Event Dates | 12 |
| 7.1.6 Conventions for Missing Concomitant Medication Dates | |
| 7.2 Analysis Sets | 12 |
| 7.3 Disposition of Subjects | 12 |
| 7.3.1 Study Information | |
| 7.3.2 Screen Failures | 13 |
| 7.3.3 Subject Eligibility | |
| 7.3.4 Number of Subjects Randomized by Site and Treatment Group | j14 |
| 7.35 Disposition of Subjects | 14 |
| 7.3.6 Protocol Deviations and Analysis Sets | 15 |
| Demographic and Other Baseline Characteristics | 16 |
| 7.5 Medical History and Concurrent Medical Conditions | 17 |
| 7.6 Medication History and Concomitant Medications | 17 |
| 7.7 Study Drug Exposure and Compliance | 18 |
| 7.8 Efficacy Analysis | 18 |

| 7.8 | .1 Primary Endpoint | 18 |
|---|---|---|
| 7.8 | .2 Secondary Endpoint | 20 |
| 7.8 | .3 Additional Efficacy Endpoint. | 20 |
| 7.8 | .4 Statistical/Analytical Issues | 21 |
| 7.9 | .4 Statistical/Analytical Issues Safety Analysis | c23 |
| 7.9 | .1 Adverse Events | 23 |
| 7.9 | .2 Clinical Laboratory Evaluations. | 26 |
| 7.9 | .3 Vital Signs and Weight | 28 |
| 7.9 | .4 12-Lead ECGs | 29 |
| 7.9 | Safety Analysis 1 Adverse Events 2 Clinical Laboratory Evaluations 3 Vital Signs and Weight 4 12-Lead ECGs 5 Other Observations Related to Safety Interim Analysis Changes in the Statistical Analysis Plan FERENCES PENDIX Criteria for Markedly Abnormal Values Criteria for Elevated Liver Enzyme Statistical Analysis Plan Version 3 Summers of Changes | 30 |
| 7.10 | Interim Analysis | 30 |
| 7.11 | Changes in the Statistical Analysis Plan. | 30 |
| 8.0 RE | FERENCES | 31 |
| 9.0 AP | PENDIX | 32 |
| 9.1 | Criteria for Markedly Abnormal Values | 32 |
| 9.2 | Criteria for Elevated Liver Enzyme | 34 |
| 9.3 | Statistical Analysis I fall version 3 Summary of Changes | 36 |
| LIST OF | IN-TEXT TABLES | |
| Table 7.a | Visit Window of <sup>13</sup> C-URP | 11 |
| Table 7.a | Visit Window of C-OBT Visit Window of Laboratory Test Values, ECG, and Vital Signs | |
| Table 7.c | Visit Window of Weight | |
| Table 9.a | MAV Criteria for Hematology | |
| Table 9.b | MAV Criteria for Serum Chemistry | |
| Table 9.c | MAV Criteria for Vital Signs | |
| Table 9.d | MAV Criteria for 12-lead ECG. | |
| Table 9.e | Criteria for Elevated Liver Enzyme. | 34 |
| 1 4010 7.0 | Official for Dievated Diver Difference | 54 |
| 1 | | |
| LIST OF | IN-TEXT FIGURES | |
| Figure 4 a | Schematic of Study Design | 7 |

#### 3.0 LIST OF ABBREVIATIONS

| <sup>13</sup> C-UBT | <sup>13</sup> C-urea breath test |
|---------------------|----------------------------------|
| CCDI | C di ca di catti test |

γ-GTP gamma-glutamyl transferase

ΑE adverse event

ALT alanine aminotransferase ALP alkaline phosphatase **AST** aspartate aminotransferase

BID twice daily **BMI** body mass index BUN blood urea nitrogen CI confidence interval CK creatine kinase

**CPK** creatine phosphokinase **ECG** electrocardiogram **FAS** full analysis set

HP Helicobacter pylori/ H.pylori lactate dehydrogenase LDH LLN lower limit of normal MAV markedly abnormal value

and subject to the applicable terms of Use applicable terms of Use Medical Dictionary for Regulatory Activities MedDRA

MIC minimum inhibitory concentration

O/E overencapsulated S PPS per protocol set preferred term PT

pretreatment adverse event PTE

catment red blood cel system organ total bilirubin treatment-emer-upper limit white 'v' system organ class

treatment-emergent adverse event

upper limit of normal white blood cell

World Health Organization

#### 4.0 **OBJECTIVES**

#### **Primary Objective** 4.1

The primary objective of this study:

To demonstrate the efficacy of HP eradication with bismuth-containing quadruple therapy with TAK-438 versus esomeprazole in all HP+ subjects.

Secondary Objects cable cert

#### 4.2 **Secondary Objectives**

Secondary objectives of this study are:

- To demonstrate the efficacy of HP eradication with bismuth-containing quadruple therapy with TAK-438 versus esomeprazole in clarithromycin resistant HP+ subjects.
- To compare the safety of bismuth-containing quadruple therapy with TAK-438 versus and subject. esomeprazole in subjects with HP infection.

#### 4.3 **Additional Objectives**

Not applicable.

#### 4.4 **Study Design**

This is a randomized, double-blind, phase 3 study to compare the efficacy and safety of bismuth-containing quadruple therapy administered with either oral TAK-438 20 mg or esomeprazole 20mg BID in all HP+ subjects?

Treatment Period—Dose and Regiment

HP+ subjects whose eligibility is confirmed will take O/E TAK-438 20 mg or O/E esomeprazole 20 mg (which are identical in appearance) BID in conjunction with bismuth-containing quadruple therapy for 2 weeks (amoxicillin 1 g BID, clarithromycin 500 mg BID, and bismuth potassium citrate 600 mg [equivalent to 220 mg bismuth], BID). The randomization ratio of TAK-438 group to esomeprazole group is 1:1.

A bacteriological test will be performed to determine if there are any resistant bacteria to the antibiotics used in the study. Biopsy specimens will be obtained from the central greater curvature of the antrum and upper greater curvature of the gastric body at the start of study (Visit 1). MICs of amoxicillin and clarithromycin against HP will be determined using the strains isolated from these specimens by the 2-fold agar dilution method. Cla >2, Amo >0.5 µg/mL is determined as resistance breakpoint.

#### Follow-up Period:

The subjects will be followed up at Week 4 post-treatment to provide a post-study <sup>13</sup>C-UBT to ascertain HP eradication status and to evaluate safety.



#### 5.0 ANALYSIS ENDPOINTS

#### Primary Endpoint

The primary endpoint for this study is the:

• Proportion of all HP+ subjects with successful HP eradication after the double-blind treatment period, as determined by <sup>13</sup>C-UBT at Week 4 post-treatment.

## Additional Endpoint

The additional endpoint for this study is the:

icable Terms of Use Librat Wand subject to the commercial use only and subject to the commercial use of the commercia • Proportion of baseline clarithromycin resistant HP+ subjects with successful HP eradication after the double-blind treatment period, as determined by <sup>13</sup>C-UBT at Week 4 post-treatment.

#### 6.0 **DETERMINATION OF SAMPLE SIZE**

This study is planned to begin with 425 randomized subjects in total (which ensures

This sample size provides over 90% power to establish noninferiority using the Farrington and Manning test with a noninferiority margin of 10% (1-sided 2.5% overall significance leading assuming that the true eradication rates are 000/ feed assuming that the true eradication rates are interim analysis is performed at 50% information fraction with critical value which is obtained from an O'Brien-Fleming type alpha spending function (2.96259 and 1.96860 for interim and Proparty of Takeda: For non-commercial use only and subject to the proparty of Takeda: For non-commercial use only and subject to the proparty of Takeda: final analysis, respectively). And, this provides approximately 80% power to establish superiority using score test, assuming that the true eradication rates are 95% for TAK-438 and

#### 7.0 METHODS OF ANALYSIS AND PRESENTATION

## 7.1 General Principles

#### 7.1.1 Study Definitions

The following definitions and calculation formulas will be used.

- Descriptive statistics: Number of subjects, mean, standard deviation, maximum, minimum, and quartiles
- BMI (kg/m<sup>2</sup>): Weight (kg) / height (m)<sup>2</sup> (rounded to 1 decimal place)
- Clarithromycin Resistant: A subject will be considered clarithromycin resistant if maximum of the MICs of clarithromycin against HP is  $>2 \mu g/mL$
- Amoxicillin Resistant: A subject will be considered amoxicillin resistant if maximum of the MICs of amoxicillin against HP is >0.5 μg/mL
- Duration of exposure to study drug (days): Date of last dose of study drug date of first dose of study drug + 1
- Study drug compliance (%) (rounded to 1 decimal place).
  - TAK-438/esomeprazole: Number of study drugs taken / 28 \* 100
  - Amoxicillin: Number of study drugs taken 56 \* 100
  - Clarithromycin: Number of study drugs taken / 56 \* 100
  - Bismuth potassium citrate: Number of study drugs taken / 56 \* 100
- TEAE: An adverse event whose date of onset occurs on or after the start of study drug. An event whose type entered into the EDC is Adverse Event will be treated as a TEAE if its start date is missing.
- PTE: Any untoward medical occurrence in a clinical investigation subject who has signed informed consent to participate in a study but prior to administration of any study drug
- Relationship of TEAE to study drug: If relationship to study drug is missing, the TEAE is considered to be a drug-related TEAE in analyses
- Intensity of TEAE: If intensity is missing, the TEAE is considered to be a severe TEAE in analyses
- Significant TEAE: Any TEAE (not including serious TEAE) that led to an intervention, including withdrawal of drug treatment, dose increase, dose reduction, dose interruption or significant additional concomitant therapy
- QTcF interval (msec): QT interval (msec) / RR interval (sec)<sup>0.33</sup> (rounded to the whole number)

#### 7.1.2 Definition of Study Days

The following definitions and calculation formulas will be used.

- Study Day: The day before the first dose of the study drug will be defined as Study Day -1 and the day of the first dose will be defined as Study Day 1.
- Follow-up Day: The day after the last dose of the study drug will be defined as Follow-up Day 1.

## 7.1.3 Definition of Study Visit Windows

When calculating Study Day relative to a reference date (i.e., date of first dose of study drug [Day 1]), if the date of the observation is on the same date or after the reference date, it will be calculated as: date of observation - reference date + 1; otherwise, it will be calculated as: date of observation - reference date. Hence, reference day is always Day 1 and there is no Day 0.

When calculating Follow-up Day relative to a reference date (i.e., date of last dose of study drug [Follow-up Day 0]), it will be calculated as: date of observation, reference date. Hence, reference day is always Follow-up Day 0.

All evaluable data (i.e., non-missing data) will be handled according to the following rules.

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Day to the scheduled Study Day will be used. If there are 2 observations equidistant to the scheduled Study Day, the later observation will be used.

Table 7.a Visit Window of <sup>13</sup>C-UBT

| Visit | Scheduled Study Day | Time Inter | val (days) |
|-----------------------|---------------------|------------|---------------|
| V ISIT | (days) | Study Day | Follow-up Day |
| Week 4 Post-Treatment | Follow-up Day: 28 | | 28 - 35 |

Table 7.b Visit Window of Laboratory Test Values, ECG, and Vital Signs

| | Visit | Scheduled Study Day | Time Inter | val (days) |
|---|------------------|---------------------|------------|---------------|
| l | VISIT O | (days) | | Follow-up Day |
| ĺ | Baseline | Study Day: 1 | -28 - 1 | |
| ı | End of Treatment | Study Day: 15 | 2 <= | <15 |

Table 7.c Visit Window of Weight

| Visit | Scheduled Study Day | Time Inter | val (days) |
|---|---|---|---|
| V 151t | (days) | Study Day Follow-up I | |
| Baseline | Study Day: 1 | -28 - 1 | |
| Week 4 Post-Treatment | Follow-up Day: 28 | | 28 - 35 |

## Significance Level and Confidence Coefficient

- Significance level: 2.5% (1-sided test)
- Confidence coefficient: 95% (2-sided)

#### **Conventions for Missing Adverse Event Dates**

Not applicable.

## **Conventions for Missing Concomitant Medication Dates**

Not applicable.

#### 7.2 **Analysis Sets**

FAS:

icable Terms of Use se of All subjects who were randomized and received at least 1 dose of study drug. Analyses based on the FAS will be performed according to the randomization assignment.

PPS:

All FAS subjects who did not have any of the major protocol deviations listed below, and whose primary endpoint was evaluable

- Subjects who did not meet inclusion criteria #4
- Subjects who met exclusion criteria #5, #6, #7, or #10
- Subjects with any of the study medication compliances of less than 70%
- Subjects who have been unblinded by the investigator prior to database lock
- Subjects who have violated the rules specified in section 7.3 of the protocol

Analyses based on the PPS will be performed according to the actual treatment received.

Safety analysis set:

All subjects who received at least 1 dose of study drug. Analyses based on the safety analysis set will be performed according to the actual treatment received.

#### 7.3 **Disposition of Subjects**

# 7.3.1 Study Information

Analysis Set:

All Subjects Who Signed the Informed Consent Form

Analysis Variables:

Date First Subject Signed Informed Consent Form

Date of Last Subject's Last Visit/Contact

MedDRA Version

WHO Drug Version

SAS Version Used for Creating the Datasets

Analytical Methods:

(1) Study Information

Study information shown in the analysis variables section will be provided.

#### 7.3.2 Screen Failures

Analysis Set:

All Subjects Who Were Not Randomized

Analysis Variables:

Gender

Analytical Methods:

(1) Screen Failures

Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided.

#### 7.3.3 **Subject Eligibility**

Analysis Set:

All Subjects Who Signed the Informed Consent Form

Analysis Variables:

Eligibility Status

[Eligible for Randomization, Not Eligible for Randomization]

Primary Reason for Subject Not Being Eligible

[Adverse Event, Protocol Deviation, Lost to Follow-up, Voluntary Withdrawal by Subject, Study Terminated by Sponsor, Screen Failure, Other]

Subje Analytical Methods:

(1) Eligibility for Randomization

Frequency distributions will be provided. When calculating percentages for the primary reasons for subject not being eligible, the total number of ineligible subjects will be used as the denominator.

## 7.3.4 Number of Subjects Randomized by Site and Treatment Group

Analysis Set:

Randomized Set

Analysis Variables:

Randomization Status

[Randomized]

Stratum:

Site [Site numbers will be used as categories]

Analytical Methods:

applicable Terms of Use (1) Number of Subjects Randomized by Site and Treatment Group

Frequency distribution will be provided for each stratum by treatment group and Set

Study Drug Administration Status

[Randomized but Not Time
Reason for Not Being [A.]

## 7.3.5 Disposition of Subjects

Analysis Set:

Analysis Variables:

[Adverse Event, Protocol Deviation, Lost to Follow-up, Voluntary Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Lack of Efficacy, Other]

Study Drug Completion Status

[Completed Study Drug, Prematurely Discontinued Study Drug]

Reason for Discontinuation of Study Drug

[Adverse Event, Protocol Deviation, Lost to Follow-up, Voluntary Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Lack of Efficacy, Other]

Completion Status of the Follow-up Period

[Completed Follow-up Period, Prematurely Discontinued Follow-up Period]

Reason for Discontinuation of the Follow-up Period

[Adverse Event, Protocol Deviation, Lost to Follow-up, Voluntary Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Lack of Efficacy, Other]

#### Analytical Methods:

#### (1) Disposition of Subjects

Frequency distributions will be provided for each treatment group and overall. When calculating percentages for the reasons for not being treated. calculating percentages for the reasons for not being treated, the total number of subjects not treated by the study drug will be used as the denominator. When calculating percentages for the reasons for discontinuation, the total number of subjects who prematurely discontinued will be used as the denominator.

## (2) Flow Diagram of Subject Disposition

A flow diagram which shows, for each treatment group, the number of subjects who were randomized, received assigned treatment, discontinued study drug with reasons, Jee Only and subject to the and discontinued follow-up period with reasons will be presented.

#### 7.3.6 **Protocol Deviations and Analysis Sets**

#### 7.3.6.1 Protocol Deviations

Analysis Set:

Randomized Set

Analysis Variables:

Significant Protocol Deviation

[Entry Criteria, Concomitant Medication, Procedure Not Performed Per Protocol, Study Medication, Withdrawal Criteria, Otherl

#### Analytical Methods:

#### (1) Protocol Deviations

Frequency distribution will be provided by treatment group and overall for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the same category will be counted only once.

7.3.6.2 Analysis Sets

Analysis Set:

Randomized Set

Analysis Variables:

**Analysis Sets** 

Full Analysis Set [Included] Per Protocol Set [Included]
Safety Analysis Set [Included]

Analytical Methods:

(1) Analysis Sets

Frequency distributions will be provided by treatment group and overall.

## 7.4 Demographic and Other Baseline Characteristics

Analysis Set:

**FAS** 

Analysis Variables:

Gender [Male, Female]

Race [American Indian or Alaska Native, Asian, Black or African American,

Native Hawaiian or Other Pacific Islander, White]

Height (cm) 
$$[Min <= -<150, 150 <= -<160, 160 <= -<170, 170 <= -<=Max]$$

Weight (kg) at Baseline

BMI (kg/m<sup>2</sup>) at Baseline

Smoking Classification

[Never Smoked, Current Smoker, Ex-Smoker]

Alcohol Consumption

[Everyday, Couple of Days Per Week, Couple of Days Per Month, Never, Former Drinker]

Caffeine Consumption [Yes, No]

Clarithromycin Resistant [Yes, No]

Amoxicillin Resistant [Yes, No]

Analytical Methods:

(1) Summary of Demographics and Baseline Characteristics

Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided by treatment group and overall.

#### 7.5 **Medical History and Concurrent Medical Conditions**

Analysis Set:

Safety Analysis Set

Analysis Variables:

Medical History

**Concurrent Medical Conditions** 

Analytical Methods:

- (1) Medical History by System Organ Class and Preferred Term
- icable Terms of Use (2) Concurrent Medical Conditions by System Organ Class and Preferred Term

Frequency distributions will be provided for each treatment group and overall. MedDRA dictionary will be used for coding. Summaries will be provided using SOC and PT, where SOC will be sorted alphabetically and PT will be sorted in decreasing frequency. A subject with multiple occurrences of medical history or concurrent medical condition within a SOC will be counted only once in that SOC. A subject with multiple occurrences of medical history or concurrent medical condition within a PT will be counted only once in that PT

#### **Medication History and Concomitant Medications** 7.6

Analysis Set:

Safety Analysis Set

Analysis Variables:

**Medication History** 

Concomitant Medications

Analytical Methods:

- (1) Medication History by Preferred Medication Name
- (2) Concomitant Medications That Started Prior to and Were Ongoing at Baseline as well as Those That Started After Baseline by Preferred Medication Name

Frequency distributions will be provided for each treatment group and overall. WHO Drug dictionary will be used for coding. Summaries will be provided using preferred medication names and sorted in decreasing frequency based on the number of reports. A subject who has been administered several medications with the same preferred medication name will be counted only once for that preferred medication name.

#### 7.7 **Study Drug Exposure and Compliance**

Analysis Set:

Safety Analysis Set

Analysis Variables:

Duration of Exposure to Study Drug (days)

$$[Min \le -<10, 10 \le -<12, 12 \le -<=14, 14 < -<=Max]$$

Study Drug Compliance (%)

TAK-438 or Esomeprazole

$$[Min \le -.. < 70.0, 70.0 \le -.. < 85.0, 85.0 \le -.. \le Max]$$

Amoxicillin

$$[Min \le -.. < 70.0, 70.0 \le -.. < 85.0, 85.0 \le -.. \le Max]$$

Clarithromycin

Bismuth Potassium Citrate

$$[Min <= - < 70.0, 70.0 <= - < 85.0, 85.0 <= - <= Max]$$
tassium Citrate
$$[Min <= - < 70.0, 70.0 <= - < 85.0, 85.0 <= - <= Max]$$

Analytical Methods:

(1) Study Drug Exposure and Compliance

Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided by treatment group and overall.

#### 7.8 **Efficacy Analysis**

The FAS will be the main analysis set used. The PPS will be used for an analysis performed secondarily on the primary endpoint in order to examine the robustness of the results.

# 7.8.1 Primary Endpoint

Analysis Set

Analysis Variables:

Proportion of all HP+ subjects with successful HP eradication after the double-blind treatment period, as determined by <sup>13</sup>C-UBT at Week 4 post-treatment

Analytical Methods:

## (1) Primary Analysis

The following analyses will be conducted using the FAS. Subjects whose HP eradication status determined by <sup>13</sup>C-UBT at Week 4 post-treatment is missing will be excluded from the analyses.

Frequency distributions of HP eradication status (Success/Failure) at Week 4 post-treatment as well as the proportion of subjects with successful HP eradication and its 2-sided 95% exact CI will be provided for each treatment group. The proportion difference between treatment groups and its 2-sided 95% Wald CI will also be provided.

Noninferiority of TAK-438 to esomeprazole will be evaluated using Farrington and Manning test with a noninferiority margin of 10%, and superiority of TAK-438 to esomeprazole will be evaluated using a score test if and only if the noninferiority test achieves statistical significance at either of the interim analysis or the final analysis. If the test for noninferiority is statistically significant at the interim analysis, no further analysis for noninferiority will be performed for statistical testing purposes.

The hypotheses to be evaluated in the noninferiority test are:

$$\begin{split} &H_0: \ p_{TAK-438} \leq p_{esomeprazole} - \delta \\ &H_A: \ p_{TAK-438} > p_{esomeprazole} - \delta \end{split}$$

and the hypotheses to be evaluated in the superiority test are:

$$H_0$$
:  $p_{TAK-438} \le p_{esome prazole}$   
 $H_A$ :  $p_{TAK-438} > p_{esome prazole}$ ,

where  $p_{TAK-438}$  and  $p_{esomeprazole}$  are the proportion of subjects with successful HP eradication at Week 4 post-treatment for TAK-438 and esomeprazole groups, respectively, and  $\delta$  is the noninferiority margin (10%).

There are 2 analyses planned in this study: 1 interim analysis and the final analysis. At the interim analysis, sample size re-estimation will also be performed based on the conditional powers for noninferiority and superiority tests. Inflation of type 1 error rate associated with multiple testing (noninferiority/superiority, interim analysis/final analysis) will be controlled using the closed testing procedure and O'Brien-Fleming type alpha spending function. Inflation of type 1 error rate associated with the sample size re-estimation will be controlled using Cui-Hung-Wang test [1] at the final analysis based on the stage-wise test statistics by Farrington and Manning test for noninferiority and score test for superiority. The actual critical values for the interim analysis and the final analysis, and the actual weights for Cui-Hung-Wang test will be determined based on the observed information fraction in the first stage and the initial sample size for the primary analysis of 400.

#### (2) Secondary Analysis

The same analyses as those in the primary analysis will be conducted using the PPS.

#### (3) Other Analysis

In order to evaluate the impact of subjects whose HP eradication status determined by <sup>13</sup>C-UBT at Week 4 post-treatment is missing, the following two types of analyses will be conducted including:

- 1) All subjects in the FAS whose HP eradication status determined by <sup>13</sup>C-UBT post-baseline is available (i.e. without applying visit window of <sup>13</sup>C-UBT in Table 7.a., and excluding subjects whose HP eradication status post-baseline is missing).
- All subjects in the FAS, where i) HP eradication status determined by <sup>13</sup>C-UBT post-baseline will be used for subjects whose HP eradication status is available post-baseline, and ii) HP eradication status will be treated as Failure for subjects whose HP eradication status post-baseline is missing.

For both of the analyses 1) and 2) above, frequency distributions of HP eradication status (Success/Failure) at Week 4 post-treatment as well as the proportion of subjects with successful HP eradication and its 2-sided 95% exact CI will be provided for each treatment group. The proportion difference between treatment groups and its 2-sided 95% Wald CI will also be provided.

# 7.8.3 Additional Efficacy Endpoint Analysis Set: FAS

Analysis Variables:

Proportion of baseline clarithromycin resistant HP+ subjects with successful HP eradication after the double-blind treatment period, as determined by <sup>13</sup>C-UBT at Week 4 post-treatment

Analytical Methods:

The following analyses will be conducted for subjects in the FAS who are clarithromycin resistant at baseline and whose HP eradication status determined by <sup>13</sup>C-UBT at Week 4 post-treatment is non-missing.

Frequency distributions of HP eradication status (Success/Failure) at Week 4 post-treatment as well as the proportion of subjects with successful HP eradication and its 2-sided 95% exact CI will be provided for each treatment group. The proportion difference between treatment groups and its 2-sided 95% Wald CI will also be provided.

#### 7.8.4 Statistical/Analytical Issues

#### 7.8.4.1 Adjustments for Covariates

Adjustments for covariates are currently not planned in this study.

#### 7.8.4.2 Handling of Dropouts or Missing Data

Missing test results will not be used for hypothesis testings and estimations unless otherwise specified.

Values below the lower limit of quantification will be treated as zero when calculating the descriptive statistics. Values greater than or equal to the upper limit of quantification will be treated as the upper limit value when calculating the descriptive statistics.

#### 7.8.4.3 Multicenter Studies

Evaluation of treatment-by-center interaction is currently not planned in this study.

#### 7.8.4.4 Multiple Comparison/Multiplicity

Two types of statistical tests are planned for the primary endpoint: noninferiority and superiority, at the interim analysis and the final analysis. Inflation of type 1 error rate associated with this multiple testing will be controlled using the closed testing procedure and O'Brien-Fleming type alpha spending function. More specifically, the superiority test of TAK-438 to esomeprazole will be performed if and only if the noninferiority test of TAK-438 to esomeprazole achieves statistical significance, and the critical values for the interim and the final analyses will be calculated based on the O'Brien-Fleming type alpha spending function. Also, inflation of type 1 error rate associated with the sample size re-estimation will be controlled using Cui-Hung-Wang test [1] at the final analysis.

# 7.8.4.5 Use of an "Efficacy Subset" of Subjects

In addition to analyses on the primary endpoint using the FAS, a secondary analysis will also be performed using the PPS to examine the robustness of the results.

# 7.8.4.6 Active-Control Studies Intended to Show Equivalence or Non-Inferiority

For the primary endpoint, noninferiority of TAK-438 to esomeprazole will be evaluated with a noninferiority margin of 10% using Farrington and Manning test as described in 7.8.1 (1) Primary Analysis.

In phase 3 studies of PPI-based triple therapy (PPI, amoxicillin and clarithromycin) in HP+ subjects, the proportions of subjects with successful HP eradication were 86.4-89.2% [2], 78.8-83.0% [3], and 85.7-91.4% [4] for lansoprazole, omeprazole, and rabeprazole, respectively, showing the variation in the results greater than 10% (78.8-91.4%).

On the other hand, very low percentage of HP eradication were observed for lansoprazole or amoxicillin monotherapy. The proportions of subjects with successful HP eradication for

lansoprazole monotherapy were 0.0% and 4.4% for subjects with gastric ulcer and duodenal ulcer, respectively, in the phase 3 study comparing lansoprazole monotherapy and lansoprazole-Furthermore, host factors, such as drug metabolism, as well as factors such as drug resistance may have some effects on HP eradication result.

For these reasons, the noninferiority many have some effects of HP eradication result. based triple therapy (lansoprazole, amoxicillin and clarithromycin) [2]. The proportions of

primary analysis of this study although limited data are available for the efficacy of PPI-based bismuth-containing quadruple therapy (PPI, amoxicillin, clarithromycin and bismuth potassium citrate).

#### 7.8.4.7 Examination of Subgroups

Analysis Set:

**FAS** 

Analysis Variables:

Proportion of all HP+ subjects with successful HP eradication after the double-blind treatment period, as determined by <sup>13</sup>C-UBT at Week 4 post-treatment

Subgroups:

[Min<=-<65, 65<= - <=Max] [Male, Female] Age (years)

Gender

[Yes, No] Clarithromycin Resistant

[Yes, No] Amoxicillin Resistant

Analytical Methods:

(1) Subgroup analysis of proportion of subjects with successful HP eradication at Week 4 post-treatment

For each subgroup, the following analyses will be conducted. Subjects whose HP eradication status determined by <sup>13</sup>C-UBT at Week 4 post-treatment is missing will be excluded from the analyses.

Frequency distributions of HP eradication status (Success/Failure) at Week 4 post-treatment as well as the proportion of subjects with successful HP eradication and its 2-sided 95% exact CI will be provided for each treatment group. The proportion difference between treatment groups and its 2-sided 95% Wald CI will also be provided.

to the applicable Terms of Use

## 7.9 Safety Analysis

#### 7.9.1 Adverse Events

7.9.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set:

Safety Analysis Set

Analysis Variables:

**TEAE** 

Categories:

Relationship to Study Drug [Related, Not Related]

Intensity [Mild, Moderate, Severe]

Analytical Methods:

The following summaries will be provided for each treatment group.

- (1) Overview of Treatment-Emergent Adverse Events
  - 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - 2) Relationship of Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
  - 3) Intensity of Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - 4) Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
  - 5) Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - 6) Relationship of serious Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
    - Serious Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
  - 8) Treatment-Emergent Adverse Events resulting in death (number of events, number and percentage of subjects)

TEAEs will be counted according to the rules below.

#### Number of subjects

• Summaries for 2) and 6)

A subject with occurrences of TEAE in both categories (i.e., Related and Not Related) will be counted once in the Related category.

• Summary for 3)

A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.

Summaries other than 2), 3), and 6)

A subject with multiple occurrences of TEAE will be counted only once.

#### Number of events

For each summary, the total number of events will be calculated. use only and subject

7.9.1.2 Displays of Treatment-Emergent Adverse events

Analysis Set:

Safety Analysis Set

Analysis Variables:

**TEAE** 

Categories:

[Mild, Moderate, Severe] Intensity

Analytical Methods:

The following summaries will be provided using frequency distribution for each treatment group.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT.

SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by SOC only or PT only.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (2) Treatment-Emergent Adverse Events by System Organ Class
- (3) Treatment-Emergent Adverse Events by Preferred Term
- (4) Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (5) Intensity of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (6) Intensity of Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (7) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term
- (8) Drug-Related Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term
- (9) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (10) Drug-Related Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (11) Significant Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (12) Most Frequent Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (13) Most Frequent Non-Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

Most frequent TEAEs refer to PTs whose percentages are at least 2% in any one of the treatment groups.

Most frequent non-serious TEAEs refer to PTs whose percentages are at least 5% in any one of the treatment groups. If there are no PTs that meet this criterion, the threshold will be lowered to 2%. The number of subjects who experienced any one of the most frequent non-serious TEAEs will also be displayed in this summary.

The frequency distribution will be provided according to the rules below.

#### Number of subjects

• Summary tables other than (5) and (6)

A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT.

Summary tables for (5) and (6)

Applicable Terms of Use A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity.

## 7.9.1.3 Displays of Pretreatment Events

#### Analysis Set:

All Subjects Who Signed the Informed Consent Form

Analysis Variables:

**PTE** 

#### Analytical Methods:

The following summaries will be provided using frequency distribution.

PTEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

- (1) Pretreatment Events by System Organ Class and Preferred Term
- (2) Serious Pretreatment Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below.

#### Number of subjects

A subject with multiple occurrences of PTE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only once in that PT.

## **Clinical Laboratory Evaluations**

## 7.9.2.1 Hematology and Serum Chemistry

Analysis Set:

Safety Analysis Set

Analysis Variables:

Hematology

Erythrocytes (RBC), Leukocytes (WBC), Hemoglobin, Hematocrit, Platelets, Neutrophils, Eosinophils, Basophils, Monocytes, Lymphocytes

## Serum Chemistry

ALT, ALP, AST, y-GTP, TB, Direct Bilirubin, LDH, CK (CPK), Albumin, Total Protein, Creatinine, BUN, Urate, Total Cholesterol, Triglycerides (Fasting), Glucose (Fasting), Potassium, Sodium, Magnesium, Calcium, Phosphate, Chloride

Visit:

Baseline, End of Treatment

## Analytical Methods:

- For applicable variables, summaries (1) and (2) will be provided by treatment group.

  (1) Summary of Laboratory Test Results and Change from Baseline by V.

  Descriptive statistics for observed. will be provided.
- (2) Summary of Shifts of Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

For each laboratory test, the laboratory values will be classified as "Low", "Normal" or "High" relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications.

(3) Number and Percentage of Subjects with Markedly Abnormal Values of Laboratory **Parameters** 

Overall frequency distributions of MAV after baseline will be provided. If a laboratory parameter has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix.

(4) Number and Percentage of Subjects with Elevated Liver Enzyme Laboratory **Parameters** 

Overall frequency distributions of elevated hepatic parameters after baseline will be provided. Further details are given in Appendix.

## 7.9.2.2 Urinalysis

Analysis Set:

Safety Analysis Set

Analysis Variables:

Protein

Glucose

Baseline, End of Treatment

Analytical Methods:

For each variable, summary (1) will be provided by treatment group.

(1) Summary of Shifts of Urine Laboratory Test Results

and subject to the applicable Terms of Use Diast Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

## 7.9.3 Vital Signs and Weight

Analysis Set:

Safety Analysis Set

Analysis Variables:

**Body Temperature** 

Systolic Blood Pressure

Diastolic Blood Pressure

Respiration Rate

Pulse Rate

Weight

Visit:

Body Temperature, Systolic Blood Pressure, Diastolic Blood Pressure, Respiration Rate, Pulse Rate:

Baseline, End of Treatment

Baseline, Week 4 Post-Treatment

Analytical Methods:

For each variable, summary (1) will be provided by treatment group.

For applicable variables, summary (2) will be provided by treatment group.

- (1) Summary of Vital Signs Parameters and Change from Baseline by Visit Descriptive statistics for observed values for each visit and changes from baseline will be provided.
- Number and Percentage of Subjects with Markedly Abnormal Values of Vital Signs Parameters

Overall frequency distributions of MAV after baseline will be provided. If a vital sign parameter has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix.

#### **7.9.4 12-Lead ECGs**

Analysis Set:

Safety Analysis Set

Analysis Variables:

Heart Rate

RR Interval

PR Interval

**QRS** Interval

QT Interval

**QTcF** Interval

Interpretation

The applicable Terms of Use by so [Within Normal Limits, Abnormal but not Clinically Significant, Abnormal and Clinically Significant]

Visit:

Baseline, End of Treatment

Analytical Methods:

For each variable other than 12-lead ECG interpretations, summary (1) will be provided by treatment group.

For applicable variables, summary (2) will be provided by treatment group.

For 12-lead ECG interpretation, summary (3) will be provided by treatment group.

- (1) Summary of ECG Parameters and Change from Baseline by Visit Descriptive statistics for observed values for each visit and changes from baseline will be provided.
- (2) Number and Percentage of Subjects with Markedly Abnormal Values of ECG **Parameters**

Overall frequency distributions of MAV after baseline will be provided. If an ECG parameter has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix.

(3) Summary of Shift of 12-lead ECG Interpretation

Shift table showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

#### 7.9.5 Other Observations Related to Safety

Not applicable.

A single interim analysis will be conducted after approximately 200 evaluable subjects in total have been assessed for the primary endpoint. Statistical analyses for the primary endpoint by socret. by score test, and calculation of conditional powers for noninferiority test and superiority test for the purpose of sample size re-estimation. The decisions taken after the interim analysis are early stopping for efficacy (noninferiority only or both noninferiority and superiority), study continuation without sample size increase, or study continuation with sample size increase.

Type 1 error rate will be controlled by O'Brien-Fleming type alpha spending function and Cui-Hung-Wang test (for final analysis only). The actual critical values for the interim analysis and the final analysis, and the actual weights for Cui-Hung-Wang test will be determined based on the observed information fraction in the first stage and initial sample size for the primary analysis of 400.

If the test for noninferiority is statistically significant at the interim analysis, no further analysis for noninferiority will be performed for statistical testing purposes.

## **Changes in the Statistical Analysis Plan**

property of Takeda. For non-commercial The analyses in the statistical analysis plan do not differ from the analyses specified in the

#### 8.0 REFERENCES

- [1] Cui, L., Hung, HMJ. and Wang, S-J. (1999). Modification of sample size in group sequential clinical trials. *Biometrics* **55**, 853-7.
- [2] Asaka, M., Sugiyama, T., Kato, M., Satoh, K., Kuwayama, H., Fukuda, Y., ... & Kobayashi, S. (2001). A multicenter, double-blind study on triple therapy with lansoprazole, amoxicillin and clarithromycin for eradication of *Helicobacter pylori* in Japanese peptic ulcer patients. Helicobacter, **6**(3), 254-261.
- [3] Kuwayama, H., Luk, G., Yoshida, S., Nakamura, T., Kubo, M., Uemura, N., ... & Nakazawa, S. (2005). Efficacy of a low-dose omeprazole-based triple-therapy regimen for *Helicobacter pylori* eradication independent of cytochrome P450 genotype. Clinical drug investigation, **25**(5), 293-305.
- [4] Kuwayama, H., Asaka, M., Sugiyama, T., Fukuda, Y., Aoyama, N., Hirai, Y., ... & Japan Rabeprazole Study Group. (2007). Rabeprazole-based eradication therapy for *Helicobacter pylori*: a large-scale study in Japan. Alimentary pharmacology & therapeutics, **25**(9), 1105-1113
- [5] Harford, W., Lanza, F., Arora, A., Graham, D., Habere M., Weissfeld, A., ... & Siepman, N. (1996). Double-blind, multicenter evaluation of lansoprazole and amoxicillin dual therapy for the cure of *Helicobacter pylori* infection. Helicobacter, 1(4), 243-250.

#### 9.0 APPENDIX

#### 9.1 Criteria for Markedly Abnormal Values

For each parameter, all evaluable data (i.e., non-missing data) obtained after baseline and up to Follow-up Day 35 will be classified as a MAV or not. The criteria in the table below will be used.

**MAV** Criteria for Hematology Table 9.a

| Parameter | MAV Criteria | |
|---------------------------------|----------------|----------------|
| 1 at ameter | Lower Criteria | Upper Criteria |
| Erythrocytes (RBC) | <0.8×LLN | Y.2×ULN |
| Leukocytes (WBC) | <0.5×LLN | >1.5×ULN |
| Hemoglobin | <0.8×LLN | >1.2×ULN |
| Hematocrit | <0.8×LLN | >1.2×ULN |
| Platelets (×10 <sup>9</sup> /L) | <75 | >600 |
| Neutrophils | <0.5×LLN | >1.5×ULN |
| Eosinophils | - 200 | >2×ULN |
| Basophils | 14.0 | >3×ULN |
| Monocytes | 06. | >2×ULN |
| Lymphocytes | <0.5×LLN | >1.5×ULN |

MAV Criteria for Serum Chemistry Table 9.b

| Parameter (1777) | MAV Criteria | |
|----------------------------|----------------|----------------|
| rarameter | Lower Criteria | Upper Criteria |
| ALT | - | >3×ULN |
| ALP | - | >3×ULN |
| AST | - | >3×ULN |
| γ-GTP | - | >3×ULN |
| TB (μmol/L) | - | >34.2 |
| Direct Bilirubin | - | >2×ULN |
| CK (CPK) | - | >5×ULN |
| Albumin (g/L) | <25 | - |
| Total Protein | <0.8×LLN | >1.2×ULN |
| Creatinine (µmol/L) | - | >177 |
| BUN (mmol/L) | - | >10.7 |
| Total Cholesterol (mmol/L) | - | >7.72 |
| Triglycerides (Fasting) | - | >2.5×ULN |
| Glucose (Fasting) (mmol/L) | <2.8 | >19.4 |

| Parameter | MAV Criteria | |
|--------------------|----------------|----------------|
| Parameter | Lower Criteria | Upper Criteria |
| Potassium (mmol/L) | <3.0 | >6.0 |
| Sodium (mmol/L) | <130 | >150 |
| Magnesium (mmol/L) | <0.5 | >1.2 |
| Calcium (mmol/L) | <1.75 | >2.88 |
| Chloride (mmol/L) | <75 | >126 |

Table 9.c MAV Criteria for Vital Signs

| Parameter | MAV Criteria | |
|---------------------------------|----------------|----------------|
| Tarameer | Lower Criteria | Upper Criteria |
| Body Temperature (°C) | <35.6 | >37.7 |
| Systolic Blood Pressure (mmHg) | <85 | >180 |
| Diastolic Blood Pressure (mmHg) | <50 | >110 |
| Pulse Rate (bpm) | <50 | >120 |

Table 9.d MAV Criteria for 12-lead ECG

| Parameter | MAV Criteria | |
|---|---|---|
| Tarameter | Lower Criteria | Upper Criteria |
| Heart Rate (bpm) | <50 | >120 |
| QT Interval (msec) | <=50 | >=460 |
| QTcF Interval (msec) | <=50 | <ul> <li>Observed value &gt;= 500, or</li> <li>Observed value &gt;= 450 and change from baseline &gt;= 30</li> </ul> |

For each parameter and subject, classifications will be made according to the conditions i) to iii) provided below. The lower and the upper criteria will be considered separately.

- i) A subject with at least one evaluable data after baseline that meets the MAV criteria will be classified as a subject with MAV.
- ii) A subject who does not meet condition i) and has at least one evaluable data after baseline that doesn't meet the MAV criteria will be considered as a subject without MAV.
- A subject who does not meet conditions i) or ii) will be excluded from the analysis of MAV for that parameter.

## 9.2 Criteria for Elevated Liver Enzyme

All evaluable data (i.e., non-missing data) obtained after baseline and up to Follow-up Day 35 will be used to determine whether each criteria for elevated liver enzyme in the table below is met or not. If there is more than one parameter that need to be considered for a criteria, parameter measurements taken on the same day will be used.

Table 9.e Criteria for Elevated Liver Enzyme

| Table 5.c Criteria for Elevated Liver Enzyme | | |
|---|---|---|
| Label | Label Criteria for Elevated Liver Enzyme | |
| Laber | (a) Elevated | (b) Not Elevated |
| ALT > 3xULN | ALT is greater than 3 times the ULN | ALT is non-missing and less than or equal to 3 times the ULN |
| ALT > 5xULN | ALT is greater than 5 times the ULN | ALT is non-missing and less than or equal to 5 times the ULN |
| ALT > 8xULN | ALT is greater than 8 times the ULN | ALT is non-missing and less than or equal to 8 times the ULN |
| ALT > 3xULN<br>with TB > 2xULN | ALT is greater than 3 times the ULN and the total bilirubin is greater than twice the ULN | Either ALT is non-missing and less than or equal to 3 times the ULN, or the total bilirubin is non-missing and less than or equal to twice the ULN |
| AST > 3xULN | AST is greater than 3 times the ULN | AST is non-missing and less than or equal to 3 times the ULN |
| AST > 5xULN | AST is greater than 5 times the ULN | AST is non-missing and less than or equal to 5 times the ULN |
| AST > 8xULN | AST is greater than 8 times the ULN | AST is non-missing and less than or equal to 8 times the ULN |
| AST > 3xULN<br>with TB > 2xULN | AST is greater than 3 times the ULN and the total bilirubin is greater than twice the ULN | Either AST is non-missing and less than or<br>equal to 3 times the ULN, or the total<br>bilirubin is non-missing and less than or<br>equal to twice the ULN |
| ALT or AST > 3xULN | Either ALT or AST is greater than 3 times the ULN | Both ALT and AST are non-missing and less than or equal to 3 times the ULN |
| ALT or AST > 5xULN | Either ALT or AST is greater than 5 times the ULN | Both ALT and AST are non-missing and less than or equal to 5 times the ULN |
| ALT or AST > 8XULN | Either ALT or AST is greater than 8 times the ULN | Both ALT and AST are non-missing and less than or equal to 8 times the ULN |
| ALT of AST > 3xULN<br>with TB > 2xULN | Either ALT or AST is greater than 3 times the ULN and the total bilirubin is greater than twice the ULN | If any of the following conditions is met: - Both ALT and AST are non-missing and less than or equal to 3 times the ULN. - Total bilirubin is non-missing and less than or equal to twice the ULN. |
| ALT and AST > 3xULN | Both ALT and AST are greater than 3 times the ULN | Either ALT is non-missing and less than or equal to 3 times the ULN, or AST is non-missing and less than or equal to 3 times the ULN |

| Label | Criteria for Elevated Liver Enzyme | |
|---|---|---|
| Label | (a) Elevated | (b) Not Elevated |
| ALT and AST > 5xULN | Both ALT and AST are greater than 5 times the ULN | Either ALT is non-missing and less than or equal to 5 times the ULN, or AST is non-missing and less than or equal to 5 times the ULN |
| ALT and AST > 8xULN | Both ALT and AST are greater than 8 times the ULN | Either ALT is non-missing and less than or<br>equal to 8 times the ULN, or AST is non-<br>missing and less than or equal to 8 times<br>the ULN |
| ALT and AST > 3xULN with TB > 2xULN | Both ALT and AST are greater than 3 times the ULN and the total bilirubin is greater than twice the ULN | If any of the following conditions is met: - ALT is non-missing and less than or equal to 3 times the ULN - AST is non-missing and less than or equal to 3 times the ULN - Total bilirubin is non-missing and less than or equal to twice the ULN |
| ALP > 3xULN | ALP is greater than 3 times the ULN | ALP is non-missing and less than or equal to 3 times the ULN |
| ALP > 3xULN<br>with ALT > 3xULN | Both ALP and ALT are greater than 3 time the ULN | Either ALP is non-missing and less than or<br>equal to 3 times the ULN, or ALT is non-<br>missing and less than or equal to 3 times<br>the ULN |
| ALP > 3xULN<br>with AST > 3xULN | Both ALP and AST are greater than 3 times the ULN | Either ALP is non-missing and less than or<br>equal to 3 times the ULN, or AST is non-<br>missing and less than or equal to 3 times<br>the ULN |

For each criteria and subject, classifications will be made according to the conditions i) to iii) provided below.

- A subject who met criteria (a) at least once after baseline will be considered to have met the criteria for elevated liver enzyme.
- ii) If condition i) is not met but if criteria (b) is met at least once after baseline, then the subject will be considered to have not met the criteria for elevated liver enzyme.
- iii) If neither i) nor ii) is met, then the subject will be excluded from the analysis for the criteria for elevated liver enzyme.

## 9.3 Statistical Analysis Plan Version 3 Summary of Changes

The changes from Statistical Analysis Plan version 2 are as follows:

- 7.1.1 Definition of TEAE was revised to address adverse events whose start date is completely or partially missing.
  - Old text: An adverse event whose date of onset occurs on or after the start of study drug
  - Revised text: An adverse event whose date of onset occurs on or after the start of study drug. An event whose type entered into the EDC is Adverse Event will be treated as a TEAE if its start date is missing.
- 7.8.1 (3) Other Analysis was added to evaluate the impact of subjects whose HP eradication status determined by 13C-UBT at Week 4 post-treatment is missing.
- 7.8.4.6 Active-Control Studies Intended to Show Equivalence or Non-Inferiority was revised to describe the rationale for the noninferiority margin used in the study.
  - Old text: For the primary endpoint, noninferiority of TAK-438 to esomeprazole will be evaluated with a noninferiority margin of 10% using Farrington and Manning test as described in 7.8.1 (1) Primary Analysis.
  - Revised text: For the primary endpoint, noninferiority of TAK-438 to esomeprazole will be evaluated with a noninferiority margin of 10% using Farrington and Manning test as described in 7.8.1 (1) Primary Analysis.

In phase 3 studies of PPI-based triple therapy (PPI, amoxicillin and clarithromycin) in HP+ subjects, the proportions of subjects with successful HP eradication were 86.4-89.2% [2], 78.8-83.0% [3], and 85.7-91.4% [4] for lansoprazole, omeprazole, and rabeprazole, respectively, showing the variation in the results greater than 10% (78.8-91.4%).

On the other hand, very low percentage of HP eradication were observed for lansoprazole or amoxicillin monotherapy. The proportions of subjects with successful HP eradication for lansoprazole monotherapy were 0.0% and 4.4% for subjects with gastric ulcer and duodenal ulcer, respectively, in the phase 3 study comparing lansoprazole monotherapy and lansoprazole-based triple therapy (lansoprazole, amoxicillin and clarithromycin) [2]. The proportions of subjects with successful HP eradication were both 0% for lansoprazole or amoxicillin monotherapy in a study evaluating lansoprazole and amoxicillin dual therapy [5].

Furthermore, host factors, such as drug metabolism, as well as factors such as drug resistance may have some effects on HP eradication result.

For these reasons, the noninferiority margin of 10% is considered appropriate and used in the primary analysis of this study although limited data are available for the efficacy of PPI-based bismuth containing quadruple therapy (PPI, amoxicillin, clarithromycin and bismuth potassium citrate).

| ELECTRONIC SIGNATURES | | |
|---|---|---|
| Signed by | Meaning of Signature | Server Date<br>(dd-MMM-yyyy HH:mm 'UTC' |
| Signed by Signed by Property of Takeda. For non- | ie <sup>c</sup> | ito the applicat |
| | se only and sulor | |
| | Minerciallise | |
| Forholis | | |
| and of takedai. | | |
| o copert. | | |